CLINICAL TRIAL: NCT04289727
Title: Skeletal Fragility in Type 1 Diabetes: Glycemic Control and Bone Strength
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mishaela Rubin, Associate Professor of Medicine, Columbia University
Other Study IDs: AAAS5630; R01DK122564 (NIH)
Record Dates: First submitted 2020-02-02; First posted 2020-02-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — am fasting Comprehensive Metabolic Panel (CMP) including liver function, HbA1c and 25OHD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Those with Type 1 Diabetes.
- Group 2: Those without Type 1 Diabetes.

SUMMARY:
The purpose of this research study is to find out how bones are affected in children and adolescents with type 1 diabetes (T1D) as compared to children and adolescents without type 1 diabetes.

DETAILED DESCRIPTION:
T1D is primarily associated with decrements in bone strength due to disrupted microarchitecture occurring during peak bone mass accrual, and this disruption arises from hyperglycemia and glycemic variability. Impaired bone development during this period likely predisposes to an increased fracture risk across the lifespan.

The investigators will compare baseline, 12 month and 24 month changes in High-resolution peripheral quantitative computed tomography/micro-finite element analysis (HR-pQCT/μFEA)-based estimates of bone strength and bone turnover by biochemical measurements in 40 T1D children at the onset of peak bone mineral accretion (n=40) versus sex and puberty-matched healthy controls (n=40). The investigators will determine relationships between changes in bone strength (including trabecular and cortical components) and measures of glycemic control and variability by continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria (T1D and Controls):

- Children within 2 years preceding the onset of the pubertal growth spurt

Inclusion Criteria (T1D participants):

- documentation of β-cell autoimmunity and need for insulin replacement

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR)< 60 ml/mim
* 25(OH)D level < 20 ng/ml.
* Celiac disease
* Autoimmune thyroid disease
* Addison's disease
* History of pathological fractures

  -- Disorders associated with altered skeletal structure or function
* Bone active drugs in past year
* Diabetes of other or unclear etiology

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 40 children and adolescents between the age of 8 to 14 years with type 1 diabetes and 40 children and adolescents between the age of 8 to 14 years without type 1 diabetes.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Change in microarchitecture by HR-pQCT | Two Years
  Measures of HRpQCT
Change in bone mineral density by Dual X-ray Absorptometry (DXA) | Two Years
  Measures of DXA

CONTACTS AND LOCATIONS:
Overall Officials: Mishaela Rubin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center-Harkness Pavillion, New York, New York, United States